CLINICAL TRIAL: NCT04621773
Title: Comparing the Live Birth Rate of Preimplantation Genetic Screening Versus Spontaneous Pregnancy in Patients With Unexplained Recurrent Pregnancy Loss
Brief Title: Live Birth Rate in Patients With Unexplained Recurrent Pregnancy Loss
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019SZ-087
Record Dates: First submitted 2020-11-05; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Recurrent Pregnancy Loss; Preimplantation Genetic Screening
Keywords: Unexplained Recurrent Pregnancy Loss; Preimplantation Genetic Screening; spontaneous pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PGS(Preimplantation Genetic Screening): patients with two times or more unexplained pregnancy loss, who wants to be pregnant via preimplantation genetic screening procedure
  Interventions: Procedure: Preimplantation Genetic Screening(exposure)
- SP(spontaneous pregnancy ): patients with two times or more unexplained pregnancy loss, who wants to be pregnant via spontaneous pregnancy.

INTERVENTIONS:
Procedure: Preimplantation Genetic Screening(exposure) — Preimplantation genetic screening (PGS) was developed in the late 1980s as an alternative to prenatal diagnosis for couples at risk of transmitting a genetic or chromosomal abnormality to their children. In embryos created through in vitro fertilisation (IVF), cells are biopsied and analysed using genetic tests such as polymerase chain reaction and fluorescent in situ hybridisation (FISH).
  Groups: PGS(Preimplantation Genetic Screening)

SUMMARY:
STUDY AIM: to study the pregnancy outcomes and offspring development of patient with Unexplained Recurrent Pregnancy Loss Treated by PGS and spontaneous pregnancy, and to compare the health economic indicators and patient satisfaction of the two modes of pregnancy, so as to better guide the clinical treatment.

DETAILED DESCRIPTION:
400 patients with two times or more unexplained pregnancy loss, who wants to be pregnant via preimplantation genetic screening procedure or spontaneous pregnancy are intended to be enrolled. They are going to divided into two groups: PGS(preimplantation genetic screening) group and SP(spontaneous pregnancy) group. The pregnancy outcomes and offspring development of those patients will be followed up by our investigators.

ELIGIBILITY:
Inclusion Criteria:

* patients with two times or more unexplained pregnancy loss(less than 24 weeks of gestational age, biochemical pregnancy excluded), who wants to be pregnant via preimplantation genetic screening procedure or spontaneous pregnancy.

Exclusion Criteria:

* anatomic abnormality of the reproductive system; endocrine metabolic disease; autoimmune related disease; chromosomal abnormalities; hydrosalpinx; cervical insufficiency.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients who seek treatment in our Recurrent Pregnancy Loss clinic.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 2 years of following up
  the rate of the birth of a living fetus

CONTACTS AND LOCATIONS:
Overall Officials: Rong Li, M.D., Study Chair — Center of Reproductive Medicine, Peking University Third Hospital
Locations (1):
- Center of Reproductive Medicine, Peking University Third Hospital, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murugappan G, Shahine LK, Perfetto CO, Hickok LR, Lathi RB. Intent to treat analysis of in vitro fertilization and preimplantation genetic screening versus expectant management in patients with recurrent pregnancy loss. Hum Reprod. 2016 Aug;31(8):1668-74. doi: 10.1093/humrep/dew135. Epub 2016 Jun 7. PMID 27278003